CLINICAL TRIAL: NCT04538196
Title: Coding and Documentation Education for General Surgery Residents
Brief Title: Coding Improvement Project: Resident Education on Documentation
Acronym: DER
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study staffing constraints
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Panos Kougias, Vascular Surgery Chief, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H-35600
Record Dates: First submitted 2020-03-16; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Resident Education
MeSH Terms: interventions — Clinical Coding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R Education (Experimental): Invervention: Resident who receives education on documentation and coding at the beginning of the surgical rotation
  Interventions: Other: Resident education on documentation and coding
- R no Education (No Intervention): Resident who does not receive information on documentation and coding at the beginning of the surgical rotation

INTERVENTIONS:
Other: Resident education on documentation and coding — Surgery residents will receive education on documentation and coding at the beginning of a particular surgical rotation vs the control group who will receive no education on documentation
  Arms: R Education

SUMMARY:
Most General Surgery program directors have expressed the necessity to educate residents on the business aspect of medicine. However, the literature review did not produce any interventional studies directly addressing coding and documentation in General Surgery Residents. The purpose of this study is to address specific coding and documentation mistakes as identified by surgery coding analysts in the surgical department. Through this examination, we hope to provide residents with the necessary tools and framework for adequate documentation throughout their surgical careers.

DETAILED DESCRIPTION:
Background:

Research has shown that residents have limited knowledge on documentation requirements. However, correct coding and documentation plays a pivotal role in today's health care system. Inadequate billing and coding in health record documentation can constitute fraud and abuse. Surgeons that are trained on proper billing and coding can be instrumental to reducing waste and increasing efficiency throughout the sphere of health care. The low quality of physician documentation has been widely recognized; however, definitive measures correcting the situation are absent. Truthfully, most residents are unaware that ICD-9 data is used for planning, reimbursement, quality rating, Medicare Conditions of Participation, JCAHO Core Measures thereby reinforcing the lack of understanding regarding the importance of such codes.Lack of education and time constraints results in poor physician documentation and as a consequence, inadequate coding leads to delayed or denied reimbursements. Several studies have shown under-billing and down-coding from resident encounters. However, no interventional studies directly addressing coding and documentation in General Surgery Residents were identified.

Purpose and objectives:

Objective 1: To educate general surgery residents on proper documentation; therefore, facilitating coding analyst efficiency by increasing processing time and employee satisfaction.

Hypothesis 1: Increasing note clarity will improve coding analyst productivity and output.

Objective 2: To ensure fair and accurate re-imbursement by appropriate translation of documentation to ICD-9 and CPT codes.

Hypothesis 2: Better reimbursement accuracy will result from an increase in precise, clear and complete medical records.

Objective 3: To increase self-efficacy in surgical trainees. Hypothesis 3: By incorporating appropriate documentation and coding techniques early on in their careers, we will observe increase in documentation confidence among residents.

Design and Procedure:

To initiate this study, surgical coding analysts at the Michael E. DeBakey Department of Veteran Affairs (MEDVAMC) will be interviewed on the most commonly encountered documenting mistakes in current practice at the surgery department. We intend to conduct a blinded randomized, control trial examining documentation entered by surgical trainees who receive no documentation education compared to trainee documentation after education. Endpoints will be measured by evaluating coding analyst quota which is defined as the number of charts translated into ICD-9 and CPT codes per day. Additionally, we will also be evaluating employee satisfaction as defined by the Maslach Burnout inventory; a well-researched validated survey. A time range of twelve months, starting from day one of a surgical rotation, will be used in each arm of the study. Trainees with no education on documentation will serve as the control group while those who recieve documentation education will make up the intervention group. Outcomes will be measured by changes in quota, and coder satisfaction as described above. Randomization: A randomized block design will be employed with each surgery rotation month as a unit of randomization. In other words, surgery trainees will be randomly assigned to the control or intervention group per rotating month. Since residents rotate through a surgical service every 30 days, randomization will be done per month.

Blinding and allocation concealment:

The random month assignment will take place in advance using a pre-sealed envelope containing the randomization arm that will be opened the day prior to the start of the next surgical trainee rotation. The coders and surgical trainees will be blinded to the group allocation. Furthermore, surgery residents rotating through a surgical rotation at the VA during an intervention month will be trained on documentation and coding on the first day of their rotation; the teaching session will be about 20 minutes with high yield information on proper documentation and coding. The content of the teaching session will be determined through interviews conducted with the coding analysts. In addition to this session, a note card will be provided to the residents stressing the importance of proper documentation as well as serving as a reference tool.

At the end of the rotation, an anonymous survey will be provided to the residents in order to assess if their documentation skills changed after the intervention. In addition, the coding analyst will also complete the Maslach Burnout inventory survey, a well-researched validated survey, to assess their employee's satisfaction in control vs intervention months. In addition, de-identified generally available data on the surgery department, such as relative value units and daily analyst quota will be collected. No identifiable provider information will be collected.

Data Collection and Analysis Coding Analyst satisfaction will be analyzed with the Maslach Burnout Inventory (MBI) provided at the end of each month. In addition, residents will be surveyed on knowledge on coding and documentation confidence pre and post intervention. Billing and documentation data from the surgical deparment will be collected. Data will be analyzed using the t-test to determine if increasing the clarity of notes increases productivity. Secondary outcomes: Coding analyst satisfaction scores and resident surveys will be analyzed among the intervention and control groups using t-test.The criteria used for statistical significance will correspond to a P= 0.05 and a confidence interval (CI) of 95%. Analysis will be performed with STATA IC 13.0 (Stata Corporation, College Station, TX)

ELIGIBILITY:
Inclusion Criteria:

1. All Surgery residents in the Baylor College of Medicine residency program rotating through a surgical rotation at the Michael E. DeBakey VA Medical Center between the months of November 2014 and November 2016.
2. Coding analysts employed in the Surgical Coding department at the Michael E. DeBakey VA Medical Center between the months of November 2014 and November 2016.

Exclusion Criteria:

1. Residents and coding analysts that do not wish to participate on the study,
2. Residents rotating through the a particular surigcal rotation more than once after being part of the intervention arm.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04-14 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Coding Analyst Quota | up to 72 weeks
  the number of charts translated into ICD-9 and CPT codes per day
Coding Analyst Satisfaction | up to 72 weeks
  This will be assessed by administering the Maslach Burnout inventory validated survey

SECONDARY OUTCOMES:
Relative Value Unit | up to 72 weeks
  RVU data reports will be generated on a monthly basis
Diagnosis Related Groups | up to 72 weeks
  DRG data reports will be generated on a monthly basis
Resident self-efficacy | up to 36 weeks
  Self-efficacy will be measured through a survey at the beginning and end of the surgical rotation

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Kougias, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Background] Yount KW, Reames BN, Kensinger CD, Boeck MA, Thompson PW, Forrester JD, Upchurch GR Jr, Gauger PG, Kron IL, Lau CL. Resident awareness of documentation requirements and reimbursement: a multi-institutional survey. Ann Thorac Surg. 2014 Mar;97(3):858-64; discussion 864. doi: 10.1016/j.athoracsur.2013.09.100. Epub 2013 Dec 4. PMID 24315406
- [Background] Fakhry SM. Billing, coding, and documentation in the critical care environment. Surg Clin North Am. 2000 Jun;80(3):1067-83. doi: 10.1016/s0039-6109(05)70114-6. PMID 10897279
- [Background] Fakhry SM, Robinson L, Hendershot K, Reines HD. Surgical residents' knowledge of documentation and coding for professional services: an opportunity for a focused educational offering. Am J Surg. 2007 Aug;194(2):263-7. doi: 10.1016/j.amjsurg.2006.11.031. PMID 17618817
- [Background] Benke JR, Lin SY, Ishman SL. Directed educational training improves coding and billing skills for residents. Int J Pediatr Otorhinolaryngol. 2013 Mar;77(3):399-401. doi: 10.1016/j.ijporl.2012.11.039. Epub 2012 Dec 29. PMID 23277302
- [Background] Russo R, Fitzgerald SP, Eveland JD, Fuchs BD, Redmon DP. Improving physician clinical documentation quality: evaluating two self-efficacy-based training programs. Health Care Manage Rev. 2013 Jan-Mar;38(1):29-39. doi: 10.1097/HMR.0b013e31824c4c61. PMID 22472728
- [Background] Lusco VC, Martinez SA, Polk HC Jr. Program directors in surgery agree that residents should be formally trained in business and practice management. Am J Surg. 2005 Jan;189(1):11-3. doi: 10.1016/j.amjsurg.2004.05.002. PMID 15701483